CLINICAL TRIAL: NCT01857856
Title: PHOspholamban RElated CArdiomyopathy STudy - Intervention (Efficacy Study of Eplerenone in Presymptomaticphospholamban R14del Carriers)
Brief Title: PHOspholamban RElated CArdiomyopathy STudy - Intervention
Acronym: i-PHORECAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.p. van den Berg, MD, PhD, professor in Cardiology (Other)
Collaborators: University Medical Center Groningen (Other); The Interuniversity Cardiology Institute of the Netherlands (Other Government); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Netherlands: CVON, CardioVascular Research Netherlands (Unknown)
Responsible Party: Sponsor-Investigator, M.p. van den Berg, MD, PhD, professor in Cardiology, MD PhD, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TCC2012007; 2013-001067-23 (EudraCT Number)
Record Dates: First submitted 2013-05-08; First posted 2013-05-20 (Estimated); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Phospholamban R14del Mutation-related Cardiomyopathy
Keywords: Phospholamban; cardiomyopathy; Eplerenone; presymptomatic
MeSH Terms: conditions — Cardiomyopathies | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No treatment (No Intervention): no medical treatment
- Eplerenone (Active Comparator): Eplerenone (Inspra, 50 mg for 3 years once daily) oral, film-coated tablet 50 mg for 3 years once daily
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — eplerenone (inspra; pfizer) one tablet (50mg standard dosis; 25mg reduced dosis) per day
  Other Names: Inspra
  Arms: Eplerenone

SUMMARY:
Phospholamban (PLN) R14del mutation carriers may develop dilated cardiomyopathy (DCM) and/or arrhythmmogenic cardiomyopathy (ACM). Analogous to other inherited cardiomyopathies, the natural course of the disease is age-related ("age-related penetrance"); after a presymptomatic phase of variable length many PLN R14del-carriers progress to overt disease, and are diagnosed with either DCM or ARVC. PLN is a regulator of the sarcoplasmic reticulum Ca2+-ATPase (SERCA2a) pump in cardiac muscle and thereby important for maintaining Ca2+ homeostasis. Cardiac fibrosis appears to be an early manifestation of disease. The investigators hypothesize that treatment of presymptomatic PLN R14del-carriers with eplerenone, which by virtue of its mineralocorticoid(aldosterone)-blocking properties is a strong antifibrotic agent, reduces disease progression and postpones onset of overt disease.

DETAILED DESCRIPTION:
In the Netherlands ≈15% of idiopathic dilated cardiomyopathy (DCM) and ≈10% arrhythmogenic right ventricular cardiomyopathy (ARVC) patients carry a single (founder) mutation in the gene encoding Phospholamban, PLN R14del. Analogous to other inherited cardiomyopathies, the natural course of the disease is age-related ("age-related penetrance"); after a presymptomatic phase of variable length many PLN R14del-carriers progress to overt disease, and are diagnosed with either DCM or ARVC. PLN is a regulator of the sarcoplasmic reticulum Ca2+-ATPase (SERCA2a) pump in cardiac muscle and thereby important for maintaining Ca2+ homeostasis. Cardiac fibrosis appears to be an early manifestation of disease. The investigators hypothesize that treatment of presymptomatic PLN R14del-carriers with eplerenone, which by virtue of its mineralocorticoid(aldosterone)-blocking properties is a strong antifibrotic agent, reduces disease progression and postpones onset of overt disease.

ELIGIBILITY:
Inclusion Criteria:

* Phospholamban (PLN) R14del mutation carriers
* Age ≥30 and ≤ 65 years
* New York Heart Association functional class ≤ 1
* LV ejection fraction ≥.45 (measured with MRI)

Exclusion Criteria:

* Palpitations necessitating treatment (at the discretion of the attending physician)
* A diagnosis of DCM (see appendix 1). Note: regional LV wall motions abnormalities are acceptable.
* A diagnosis of ARVC (according to the task force criteria, see appendix 2)
* Global or regional RV dysfunction and/or structural alterations (according to task force criterion 1, see appendix 2).
* Ventricular premature complexes >1000 during 24hours Holter-monitoring
* Non-sustained ventricular tachycardia during Holter-monitoring or exercise-testing
* History of sustained ventricular tachycardia or ventricular fibrillation
* Hypertension requiring the use of antihypertensive drugs, or when this is anticipated within the coming 3 years
* Evidence of ischemic heart disease
* Treatment with cardioactive medication
* Hyperkaliemia (serum potassium >5.0 mmol/l)
* Severe renal dysfunction (eGFR <30 ml/min/1.73 m2)
* Severe hepatic impairment (Child-Pugh class C)
* Women who are currently pregnant or report a recent pregnancy (last 60 days) or plan on becoming pregnant.
* Concomitant use of CYP3A4-inhibitors (see appendix 5)
* Concomitant use of NSAIDs (see appendix 5)
* Concomitant use of potassium sparing-agents (see appendix 5)
* Known intolerance or contraindication to aldosterone antagonists
* Participation in another drug trial in which the last dose of drug was within the past 30 days.
* Contra-indications for MRI (claustrophobia, metal devices)
* Subjects unable or unwilling to provide written informed consent

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2013-05; Primary Completion 2021-10 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
Left ventricular (LV) enddiastolic volume, increase >10%, as measured by MRI | three years
LV ejection fraction, absolute decrease >5%, as measured by MRI | three years
Right ventricular (RV) enddiastolic volume, increase >10%, as measured by MRI | three years
RV ejection fraction, absolute decrease >5%, as measured by MRI | three years
late gadolinium enhancement, absolute increase >5%, as measured by MRI | three years
Change in ventricular premature complexes, increase >100% in combination with absolute number >1000/24 hrs (Holter monitoring) | yearly at 0, 1, 2 and 3 years
Change in the occurrence of non-sustained ventricular tachycardia (Holter monitoring, exercise testing) | yearly at 0, 1, 2 and 3 years
Change in QRS voltage, decrease >25% (ECG) | yearly at 0,1,2 and 3 years
Change in symptoms/signs of heart failure and/or arrhythmias necessitating treatment according to the attending physician and likely due to arrhythmogenic cardiomyopathy | yearly at 0,1,2 and 3 years, and possibly in between at referral
(Change in) cardiovascular death, including sudden death, likely due to arrhythmogenic cardiomyopathy | yearly at 0,1,2 and 3 years, and possibly in between at referral

SECONDARY OUTCOMES:
Change in biomarkers | yearly at 0, 1, 2 and 3 years
Change in QRS-axis on 12-lead ECG | yearly at 0,1, 2 and 3 years
Change in conduction intervals (PR-interval, QRS-duration) on 12-lead ECG and signal averaged-ECG | yearly at 0,1, 2 and 3 years
Change in STT-segment on 12-lead ECG | yearly at 0,1, 2 and 3 years
Development of global or regional dysfunction and structural alterations on MRI | three years
(Change in) Diagnosis of ARVC (according to task force criteria) | yearly at 0,1,2 and 3 years, and possibly in between at referral
(Change in) Diagnosis of DCM | yearly at 0,1,2 and 3 years, and possibly in between at referral
Change in occurrence of sustained ventricular tachycardia or ventricular fibrillation | yearly at 0,1,2 and 3 years, and possibly in between at referral
(Change in) hospitalization for a cardiovascular reason | yearly at 0,1,2 and 3 years, and possibly in between at referral

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van den Berg, MD PhD, Principal Investigator — UMCG, Department of Cardiology
Locations (4):
- Netherlands (4):
  - AMC, Amsterdam, North Holland
  - Antonius ziekenhuis Sneek, Sneek, Provincie Friesland
  - UMCG, Groningen
  - UMCU, Utrecht

REFERENCES:
- [Background] van der Zwaag PA, van Rijsingen IA, Asimaki A, Jongbloed JD, van Veldhuisen DJ, Wiesfeld AC, Cox MG, van Lochem LT, de Boer RA, Hofstra RM, Christiaans I, van Spaendonck-Zwarts KY, Lekanne dit Deprez RH, Judge DP, Calkins H, Suurmeijer AJ, Hauer RN, Saffitz JE, Wilde AA, van den Berg MP, van Tintelen JP. Phospholamban R14del mutation in patients diagnosed with dilated cardiomyopathy or arrhythmogenic right ventricular cardiomyopathy: evidence supporting the concept of arrhythmogenic cardiomyopathy. Eur J Heart Fail. 2012 Nov;14(11):1199-207. doi: 10.1093/eurjhf/hfs119. Epub 2012 Jul 20. PMID 22820313
- [Background] van Rijsingen IA, van der Zwaag PA, Groeneweg JA, Nannenberg EA, Jongbloed JD, Zwinderman AH, Pinto YM, Dit Deprez RH, Post JG, Tan HL, de Boer RA, Hauer RN, Christiaans I, van den Berg MP, van Tintelen JP, Wilde AA. Outcome in phospholamban R14del carriers: results of a large multicentre cohort study. Circ Cardiovasc Genet. 2014 Aug;7(4):455-65. doi: 10.1161/CIRCGENETICS.113.000374. Epub 2014 Jun 8. PMID 24909667
- [Background] Te Rijdt WP, Ten Sande JN, Gorter TM, van der Zwaag PA, van Rijsingen IA, Boekholdt SM, van Tintelen JP, van Haelst PL, Planken RN, de Boer RA, Suurmeijer AJH, van Veldhuisen DJ, Wilde AAM, Willems TP, van Dessel PFHM, van den Berg MP. Myocardial fibrosis as an early feature in phospholamban p.Arg14del mutation carriers: phenotypic insights from cardiovascular magnetic resonance imaging. Eur Heart J Cardiovasc Imaging. 2019 Jan 1;20(1):92-100. doi: 10.1093/ehjci/jey047. PMID 29635323
- [Background] Te Rijdt WP, van Tintelen JP, Vink A, van der Wal AC, de Boer RA, van den Berg MP, Suurmeijer AJ. Phospholamban p.Arg14del cardiomyopathy is characterized by phospholamban aggregates, aggresomes, and autophagic degradation. Histopathology. 2016 Oct;69(4):542-50. doi: 10.1111/his.12963. Epub 2016 May 12. PMID 26970417
- [Background] Te Rijdt WP, van der Klooster ZJ, Hoorntje ET, Jongbloed JDH, van der Zwaag PA, Asselbergs FW, Dooijes D, de Boer RA, van Tintelen JP, van den Berg MP, Vink A, Suurmeijer AJH. Phospholamban immunostaining is a highly sensitive and specific method for diagnosing phospholamban p.Arg14del cardiomyopathy. Cardiovasc Pathol. 2017 Sep-Oct;30:23-26. doi: 10.1016/j.carpath.2017.05.004. Epub 2017 May 30. PMID 28759816
- [Background] Te Rijdt WP, Asimaki A, Jongbloed JDH, Hoorntje ET, Lazzarini E, van der Zwaag PA, de Boer RA, van Tintelen JP, Saffitz JE, van den Berg MP, Suurmeijer AJH. Distinct molecular signature of phospholamban p.Arg14del arrhythmogenic cardiomyopathy. Cardiovasc Pathol. 2019 May-Jun;40:2-6. doi: 10.1016/j.carpath.2018.12.006. Epub 2018 Dec 21. PMID 30763825
- [Derived] Te Rijdt WP, Hoorntje ET, de Brouwer R, Oomen A, Amin A, van der Heijden JF, Karper JC, Westenbrink BD, Sillje HHW, Te Riele ASJM, Wiesfeld ACP, van Gelder IC, Willems TP, van der Zwaag PA, van Tintelen JP, Hillege JH, Tan HL, van Veldhuisen DJ, Asselbergs FW, de Boer RA, Wilde AAM, van den Berg MP. Rationale and design of the PHOspholamban RElated CArdiomyopathy intervention STudy (i-PHORECAST). Neth Heart J. 2022 Feb;30(2):84-95. doi: 10.1007/s12471-021-01584-5. Epub 2021 Jun 18. PMID 34143416